CLINICAL TRIAL: NCT06742671
Title: Performance of a Fast-track Pathway for Giant Cell Arteritis Diagnosis
Acronym: QuickDx-GCA
Status: Recruiting | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Other Study IDs: P02/043
Record Dates: First submitted 2024-12-13; First posted 2024-12-19 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: diagnostic test; ultrasonography, Doppler, color; temporal arteries, biopsy; fast track clinic
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient suspected of Giant Cell Arteritis: Patient over 50 years old suspected of Giant Cell Arteritis and presenting at least one of the following signs:
  Visual symptoms
  * Transient vision loss (amaurosis)
  * Anterior or posterior ischemic optic neuropathy
  * Occlusion of the central retinal artery and/or its branches
  * Diplopia due to paralysis of the oculomotor muscles
  * Ocular ischemic syndrome
  Suggestive signs and symptoms:
  * Recent headaches < 4 months
  * Jaw claudication
  * Scalp tenderness
  * Abnormal temporal artery examination - beaded appearance, prominence, widening, tenderness
  * Elevated C-reactive protein ≥ 10 mg/l
  Systemic symptoms:
  * Fever
  * Anemia
  * Upper limb claudication
  * Polymyalgia rheumatica Suggestive imaging result
  * Positive positron emission computed tomography scan
  * CT scan aortitis

SUMMARY:
Giant cell arteritis is a vasculitis, i.e. inflammation of the artery walls, which generally affects people over the age of 50. Diagnosis can be long and difficult, as the clinical signs are not specific (headache, pain in the jaw, scalp, shoulders and/or pelvis, abdominal pain, weight loss, etc.), but it must be made quickly, given the risk of complications.

The reference method for diagnosis was initially based on clinical suspicion and analysis of a "piece of temporal artery" (biopsy) performed in the operating theatre under local anaesthetic. Since the mid-1990s, improvements in ultrasound techniques have made it possible to identify a sign, known as a halo, on the temporal arteries that is typical of patients with Giant Cell Arteritis. A prospective multicenter study published in 2024 demonstrated that, in patients with a clinical suspicion of Giant Cell Arteritis, if a halo was found on both temporal arteries by ultrasound, there was no need for a biopsy. This study is at the origin of a change in practices in the diagnosis and care of patients suffering from this disabling disease.

To facilitate early diagnosis, a fast-track pathway has been set up. The aim is to make a rapid diagnosis, thereby reducing the risk of after-effects, shortening the length of hospital stays, considering outpatient treatment and limiting the number of biopsies.

The investigators propose to evaluate the performance of this fast-track pathway.

DETAILED DESCRIPTION:
Giant Cell Arteritis (GCA) or temporal arteritis is a systemic vasculitis (inflammation of the artery walls) that generally affects people over 50 years old, with a peak frequency between 70 and 80 years. The diagnosis is sometimes long and difficult to make due to non-specific clinical signs but must be rapid because of the risk of arterial occlusion that can lead to vision loss or stroke.

Two GCA presentations can be detected :

* an aortic form, i.e. inflammation of the aorta with specific clinical signs (abdominal pain, weight loss, ...)
* a cephalic form with unusual headaches, jaw pain, scalp pain, shoulder and/or pelvic girdle pain, and inflammatory biological signs.

The reference method for diagnosis has been based on clinical presumption. The presence of an inflammatory syndrome in biology and the analysis of a temporal artery biopsy.

Since the mid-1990s, the improvement of ultrasound techniques, particularly with the appearance of high frequency probes, made it possible to detect inflammation of the temporal arteries in some cases. Each center published retrospective studies with the aim of avoiding biopsy but without really allowing the modification of clinical practices.

A prospective multicenter study (doi: 10.7326/M23-3417) published in 2024 proved that in patients with high clinical probability of GCA, in case of bilateral positivity on temporal artery ultrasound (hypoechoic halo) it was not necessary to resort to a biopsy.

When the ultrasound of bilateral arteries (particularly temporal and axillary) showed an abnormality such as a halo (inflammation), the diagnosis was made and did not require a biopsy.

When the ultrasound was negative (or only present on one artery or another arterial axis), biopsy was necessary. In 50% of cases, the biopsy result was negative. Among these negative cases, a certain number were nevertheless retained as Giant Cell Arteritis, according to the clinician's assessment, and others were subjected to differential diagnoses.

While with a biopsy the time to perform the procedure and obtain its interpretation was 10 days, ultrasound only requires one day to make a diagnosis.

This study is at the origin of a change in diagnosing and treating patients with this Giant Cell Arteritis.

In order to facilitate early diagnosis, a fast-track pathway has been set up based on the model published in 2024 (doi: 10.26635/6965.6376).

The investigators propose to evaluate the performance of this fast-track clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patient suspected of GCA

Exclusion Criteria:

* Opposition to the use of their data

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from North Charente-Martime with suspicion of GCA that are sent to la Rochelle hospital for fast track diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Performance of the Fast Track Clinic for GCA diagnosis | From initial GCA suspicion by the clinician to the ultrasound result (up to day 7)
  Number of patients for whom the delay between GCA suspicion and ultrasound result is less than 7 days

SECONDARY OUTCOMES:
Delay in starting corticosteroids | From initial GCA suspicion by the clinician to corticosteroid prescription (up to 1 month)
  The duration between suspicion of GCA and corticosteroid prescription
Patients with an alternative diagnosis | From clinical suspicion to the final diagnosis (around 1 month)
  Number of patients with an alternative diagnosis
Patients ultrasound negative and pathology positive | From clinical suspicion to pathology results (up to 15 days)
  The number of ultrasound negative patients with a positive result according to pathology analysis of temporal artery biopsy
GCA patients with negative ultrasound and pathology | From clinical suspicion to final diagnosis (around 1 month)
  Number of patients for whom Doppler ultrasound and biopsy analysis results are negative but who are considered to have GCA by the clinician

CONTACTS AND LOCATIONS:
Overall Officials: Christophe RONCATO, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (1):
- Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the study will be shared after deidentification.
  Study protocol and statistical analysis plan will be available. Data will be available immediately following publication. Researchers who provide a methodologically sound proposal will have access to the data.
  Data will be available at www.recherche.data.gouv.fr
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] van Dantzig P, White D, Kurz J, Ming C, Kamalaksha S, Quincey V. Performance of a fast-track pathway for giant cell arteritis in Waikato, Aotearoa New Zealand. N Z Med J. 2024 Mar 22;137(1592):31-42. doi: 10.26635/6965.6376. PMID 38513202
- [Background] Denis G, Espitia O, Allix-Beguec C, Dieval C, Lorcerie F, Gombert B, Pouget-Abadie X, Toquet C, Agard C, Raimbeau A, Gautier G, Goujon JM, Durand G, Thollot-Karolewicz C, Lormeau C, Grados A, Grenot-Mercier A, El-Khoury R, Riche A, Hospital F, Visee S, Auriault ML, Landron C, Martin M, Roncato C. Diagnostic Strategy Using Color Doppler Ultrasound of Temporal Arteries in Patients With High Clinical Suspicion of Giant Cell Arteritis : A Prospective Cohort Study. Ann Intern Med. 2024 Jun;177(6):729-737. doi: 10.7326/M23-3417. Epub 2024 May 7. PMID 38710093